CLINICAL TRIAL: NCT06456281
Title: Development and Validation of Multi-omics Model for Screening of Pancreatic Cancer Using cfDNA
Brief Title: Multi-omics Model for Pancreatic Cancer Screening Using cfDNA
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Nanjing Simcere Medical Laboratory Science Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Xian-Jun Yu, Chair of Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Fudan University
Other Study IDs: P04UR086-PAAD
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer arm: Participants with new diagnosis of pancreatic cancer.
  Interventions: Diagnostic Test: A noninvasive cfDNA multi-omics assay
- Precancerous lesions arm: Participants with precancerous lesions.
  Interventions: Diagnostic Test: A noninvasive cfDNA multi-omics assay
- Healthy individuals arm: Healthy individuals without findings of clinical significance during routine health checkups.
  Interventions: Diagnostic Test: A noninvasive cfDNA multi-omics assay

INTERVENTIONS:
Diagnostic Test: A noninvasive cfDNA multi-omics assay — Peripheral venous blood samples will be collected from pancreatic cancer patients, individuals with precancerous lesions, and healthy controls. Subsequently, cfDNA will be extracted and subjected to low-pass whole genome sequencing (LP-WGS) and hybrid capture-based targeted methylation sequencing (TMS).

SUMMARY:
This is a prospective case-control study, aiming at developing a cell free DNA (cfDNA) multi-omics precise diagnostic model for screening of pancreatic cancer.

DETAILED DESCRIPTION:
Peripheral blood samples from participants with new diagnosis of pancreatic cancers, precancerous lesions and healthy individuals will be collected to characterize the cancer-specific signatures by low-pass whole-genome sequencing and target methylation sequencing using cfDNA. An ensemble multi-omics model will be trained aided by machine learning algorithm and validated in test set. The performance of this multi-omics model distinguishing pancreatic cancer from non-cancer will be evaluated.

ELIGIBILITY:
Cancer Arm

Inclusion Criteria:

* 18-75 years old
* Clinically and/or pathologically diagnosed pancreatic cancer
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures
* Physical status score ECOG 0-1

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection or febrile illness within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Precancerous Lesions Arm

Inclusion Criteria:

* 18-75 years old
* Diagnosed with pancreatic intraepithelial tumor pancreatic intraepithelial lesions (PanINs), Intraductal papillary mucinous neoplasms (IPMN) or mucinous cystic neoplasms (MCN) by radiographical assess
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection or febrile illness within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Healthy Individuals Arm

Inclusion Criteria:

* 18-75 years old
* Clinically and/or pathologically diagnosed pancreatic non-malignant disease (pancreatic intraepithelial neoplasia, pancreatic cyst and chronic pancreatitis)
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection or febrile illness within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed pancreatic cancer or precancerous lesions and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Performance of cfDNA multi-omics model for discriminating pancreatic cancer versus healthy individuals. | 12 months
  The area under the curve (AUC), sensitivity and specificity of cfDNA multi-omics model.

SECONDARY OUTCOMES:
Performance of cfDNA multi-omics model for discriminating patients with pancreatic cancer and precancerous lesions versus healthy individuals. | 12 months
  Sensitivity of cfDNA multi-omics model at specificity of 95% for discriminating patients with pancreatic cancer and precancerous lesions versus healthy individuals.
Performance of cfDNA multi-omics model for discriminating precancerous lesions versus healthy individuals. | 12 months
  Sensitivity of cfDNA multi-omics model for discriminating precancerous lesions versus healthy individuals.
Performance of pre-defined model in clinical sub-groups of interest. | 12 months
  Sensitivity of cfDNA multi-omics model for pancreatic cancer at different stages or in different pathological subtypes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University; 270 Dong An Road, Shanghai 200032, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No